CLINICAL TRIAL: NCT03380403
Title: A Clinical Trial Testing the Efficacy of PDT in Preventing Amputation in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, João Paulo Tardivo, Principal Investigator, Faculdade de Medicina do ABC
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Faculdade de medicina do ABC
Record Dates: First submitted 2017-11-24; First posted 2017-12-21 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Foot Infection; Osteomyelitis; Photo Antimicrobial Chemotherapy
Keywords: diabetic foot; Osteomyelitis; PACT; PDT; Singlet oxygen; antimicrobial; diabetes; Wagner scale
MeSH Terms: conditions — Osteomyelitis; Diabetic Foot; Diabetes Mellitus | interventions — 1-phenyl-3,3-dimethyltriazene; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: non-randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDT (Active Comparator): Methylene blue and Photon Irradiation , every each week, until total ulcer healing.
  Interventions: Radiation: PDT
- Ciprofloxacin (Active Comparator): Diabetic foot patients were treated on conventional way, using antibiotics and surgery.
  Interventions: Other: Ciprofloxacin

INTERVENTIONS:
Radiation: PDT — clinical treatment of infected diabetic foot
  Other Names: photoantimicrobial chemotherapy
  Arms: PDT
Other: Ciprofloxacin — antibiotics and or surgical debridment
  Other Names: Conventional treatment
  Arms: Ciprofloxacin

SUMMARY:
The feet of diabetic patients continue to be an important problem in medicine. In general, patients with diabetic foot have some sort of amputation, especially in underserved populations. It is clearly necessary to develop novel treatment strategies for this worldwide health problem. Photodynamic therapy (PDT) , is a low cost and highly effective alternative treatment concerning infections avoiding amputations in the diabetic foot.

DETAILED DESCRIPTION:
Patients with infected diabetic foot were grouped according to the Wagner system for classifying foot lesions. All patients presented Wagner Grade 3 classification, with osteomyelitis in one or more toes. The study included only patients who had circulatory viability.

For PDT treatment the fistula and/or ulcer was used as a gateway to the bone. The treated area (bones and fingers) was irrigated with a solution of phenothiazinium salts. After that, light irradiation was performed with optical fibers or led device above the wound. PDT treatment always in outpatients, once or twice a week.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* diabetes
* diabetic foot
* Wagner grade III

Exclusion Criteria:

* age < 18 years old
* non-diabetic
* Wagner IV and V
* ischemia

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

PRIMARY OUTCOMES:
Infection control | every month until three months , when blood count- leucocytes reach the standard value.
  blood count - leucocytes for infection

SECONDARY OUTCOMES:
Osteomyelitis evaluation | once a month, until three months, when X-ray shows bone reconstitution .
  Radiographs were used when patients presented osteomyelitis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wainwright M, Maisch T, Nonell S, Plaetzer K, Almeida A, Tegos GP, Hamblin MR. Photoantimicrobials-are we afraid of the light? Lancet Infect Dis. 2017 Feb;17(2):e49-e55. doi: 10.1016/S1473-3099(16)30268-7. Epub 2016 Nov 22. PMID 27884621
- [Background] Tardivo JP, Baptista MS, Correa JA, Adami F, Pinhal MA. Development of the Tardivo Algorithm to Predict Amputation Risk of Diabetic Foot. PLoS One. 2015 Aug 17;10(8):e0135707. doi: 10.1371/journal.pone.0135707. eCollection 2015. PMID 26281044
- [Result] Abrahamse H, Hamblin MR. New photosensitizers for photodynamic therapy. Biochem J. 2016 Feb 15;473(4):347-64. doi: 10.1042/BJ20150942. PMID 26862179
- [Result] Sahu K, Sharma M, Dube A, Gupta PK. Topical antimicrobial photodynamic therapy improves angiogenesis in wounds of diabetic mice. Lasers Med Sci. 2015 Sep;30(7):1923-9. doi: 10.1007/s10103-015-1784-8. Epub 2015 Jul 10. PMID 26160556